CLINICAL TRIAL: NCT00962689
Title: Improving Patient Care Via Proteomics Based, Microbe-Specific Detection of Chronic Rhinosinusitis
Brief Title: Clinical Study to Improve Diagnosis and Treatment of Sinusitis
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2009H0067; KL2RR025754 (NIH)
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Chronic Sinusitis
Keywords: chronic rhinosinusitis; biofilm; sinus tissue; nasal secretions; proteomics; diagnosis; decreased antibiotics; Develop a test to identify patients with sinusitis subtypes
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood nasal secretions nasal mucosa nasal polyps
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Rhinosinusitis: Patients with chronic rhinosinusitis as defined by American Academy of Otolaryngology-Head and Neck Surgery and American Rhinologic Society guidelines
- Control Group: Patients undergoing endoscopic sinus surgery for diseases other than chronic rhinosinusitis (i.e., access to pituitary gland, etc)

SUMMARY:
Chronic rhinosinusitis (CRS) is the most common chronic medical condition that affects Americans between 18-44 years of age. While significant advances have been made in the understanding of the molecular pathogenesis underlying many subtypes of CRS, this has not translated into widespread changes in how physicians manage adult or pediatric CRS. The focus of this study is intended to develop testing methods to improve the objectivity and specificity of diagnosis and allow for individualized therapy with less invasive, customized treatments instead of the traditional, empiric based, and radically exenterative therapies commonly employed in clinical practice. Specifically, it is now known that many patients with CRS have a greater concentration of non-typeable Haemophilus influenzae (NTHI) in the bacterial biofilms located within their sinus cavities compared to healthy patients. The specific hypothesis behind the proposed research is that the presence of NTHI biofilms, which are known to be highly recalcitrant, are positively correlated with the development of CRS and that unique lipooligosaccharides and inflammatory byproducts obtained from nasopharyngeal lavage fluids and/or swabs of sinus secretions may be used as a non-invasive biomarker for CRS. As a result, patients with symptoms of CRS specifically associated with NTHI biofilms could possibly obtain a non-invasive test in the physician's office that would allow the clinician to make a more accurate diagnosis and objectively follow each patient's responsiveness to customized therapy.

DETAILED DESCRIPTION:
Specific Aims:

Specific Aim 1 will test the hypothesis that a high throughput proteomics-based assay of nasopharyngeal lavage fluids and/or swabs of human sinus drainage material will be able to identify, with a high degree of sensitivity and specificity, patients with CRS specifically due to the presence of NTHI biofilms.

Specific Aim 2 will test the hypothesis that a priori assay for increased presence of phosphorylcholine-rich lipooligosaccharides in nasopharyngeal lavage fluids from chinchillas co-infected with adenovirus and biofilm forming NTHI will successfully predict, with a high degree of sensitivity and specificity, the development of CRS in this in vivo model.

Results from this project may: enable the design and conduct of a clinical trial to preoperatively identify patients with CRS earlier in their disease course (possibly prior to the initiation of long courses of empiric antibiotic therapy); aid in the development of non-surgical therapies to eradicate bacterial biofilms with the sinus cavities; result in the identification of an objective biomarker to monitor success with therapies; and ultimately lead to less morbidity and risk for complications compared to conventional surgical therapy. In addition, transforming this paradigm would make progress towards achieving the goals of the U.S. Department Health and Human Services Healthy People 2010 objective 14-19, which is "reducing the number of courses of antibiotics prescribed for the sole diagnosis of the common cold."

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic sinusitis
* Undergoing surgery for treatment of their disease

Exclusion Criteria:

* None

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from age 5 to 90 undergoing endoscopic sinus surgery for treatment of chronic rhinosinusitis
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subinoy Das, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Das S, Maeso PA, Becker AM, Prosser JD, Adam BL, Kountakis SE. Proteomics blood testing to distinguish chronic rhinosinusitis subtypes. Laryngoscope. 2008 Dec;118(12):2231-4. doi: 10.1097/MLG.0b013e318182f7f4. PMID 18978510